CLINICAL TRIAL: NCT02890121
Title: Molecular Reclassification to Find Clinically Useful Biomarkers for Systemic Autoimmune Diseases: Cross Sectional Cohort
Brief Title: Molecular Reclassification to Find Clinically Useful Biomarkers for Systemic Autoimmune Diseases:
Acronym: PRECISESADS
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: UCB Biopharma S.P.R.L. (Industry); Atrys Health (Industry); National Research Council, Spain (Other Government); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Servicio Cántabro de Salud (Other); August Pi Sunyer Biomedical Research Institute (Other); Karolinska Institutet (Other); KU Leuven (Other); Klinikum der Universität Köln (Other); Hannover Medical School (Other); Medical University of Vienna (Other); Quartz Bio S.A. (Other); Andaluz Health Service (Other Government); The Cyprus Foundation for Muscular Dystrophy Research (Other); Universidad de Granada (Other); University of Milan (Other); Université Catholique de Louvain (Other); University Hospital, Brest (Other); University of Geneva, Switzerland (Other); Szeged University (Other); Bayer (Industry); Institut de Recherches Internationales Servier (Other); Sanofi (Industry); Eli Lilly and Company (Industry); Charite University, Berlin, Germany (Other); Centro Hospitalar do Porto (Other); Institut d'Investigació Biomèdica de Bellvitge (Other); Innovative Medicines Initiative (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: PRECISESADS CS (RB 14.106)
Record Dates: First submitted 2016-08-22; First posted 2016-09-07 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Systemic Autoimmune Diseases
Keywords: SADs; Molecular Reclassification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Connective tissue diseases (CTD) or systemic autoimmune diseases (SADs) as they are known today are a group of chronic inflammatory conditions with autoimmune aetiology with few treatment options and difficult diagnosis.Brest team contribute to perform a new classification of the following systemic autoimmune diseases in a European Union's Seventh Framework Programme. The aim of this research is to reclassify the individuals affected by SADs into molecular clusters instead of clinical entities through the determination of molecular profiles using several "Omics" techniques.

DETAILED DESCRIPTION:
The main objective of the PRECISESADS project is to reclassify the individuals affected by SADs into molecular clusters instead of clinical entities through the determination of molecular profiles using several "-omics" techniques.

The specific objectives of this cross sectional study and sub-study are:

1. To identify a systemic taxonomy for patients with SADs by producing the following data in individuals with SADs and controls: genetic, epigenomic, transcriptomic, flow cytometric (from peripheral blood mononuclear and polymorphonuclear cells (PBMCs)), metabolomics and proteomic in plasma and urine, exosome analysis, classical serology (antibodies and autoantibodies), and clinical data.
2. To better characterize individual SADs at the omics level.
3. To perform clustering analyses to determine the groups of individuals who, differentially from other groups, share specific molecular features (precision medicine).
4. To identify gene expression, methylation profiles through deconvolution methods comparing a mixture of cells with subpopulations determined by flow cytometry with separated cells, cytokine profiles and plasma metabolomics using Mass Spectrometry, in a substudy of 288 individuals.

The clustering process will be data-driven with the aim to find the most homogenous and differentiated clusters of diseases that clearly separate individuals on the basis of, serological, genetic, epigenomic, cellular (cell proportions), metabolomic, proteomic (cytokines, autoantibodies) and transcriptome characteristics and differentiate them from controls and other patient clusters.

A total of 2000 patients and 666 controls will be included in the study, adjusted to the following distribution:

* A total of 400 patients diagnosed with systemic lupus erythematosus (SLE)
* A total of 400 patients diagnosed with rheumatoid arthritis (RA)
* A total of 400 patients diagnosed of scleroderma or systemic sclerosis (SSc)
* A total of 400 patients diagnosed of Sjögren's syndrome (SjS)
* A total of 400 patients diagnosed of primary antiphospholipid syndrome (PAPS) or Mixed Connective Tissue Disease (MCTD) or with undifferentiated disease • All patients will be recruited from 18 sites in Europe (Austria, Belgium, France, Germany, Italy, Portugal, Spain, Hungary and Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* · Aged 18 years or older at the time of consent

  * Diagnosed according to prevailing criteria for one of the following systemic autoimmune diseases (see Annex 2)

    * Rheumatoid arthritis (RA)
    * Scleroderma or systemic sclerosis (SSc)
    * Primary Sjögren's syndrome (SjS)
    * Systemic lupus erythematosus (SLE)
    * Primary antiphospholipid syndrome (PAPS)
    * Mixed Connective Tissue Disease (MCTD)
    * Patients with undifferentiated connective tissue disease (UCTD) for over 1 year and that do not fulfill the diagnosis of any of the above diseases.
  * Signed the informed consent form

Exclusion Criteria:

* · Patients unable to understand the procedures related to the protocol should not be included. The study is voluntary and patients must be able to give their informed consent.

  * Pregnant women
  * Neonatal lupus
  * Drug-induced lupus
  * Patients whose condition is so serious that they cannot take part in the study
  * Severe nephrotic syndrome with proteinuria >=3,5 g/day
  * Patients with stable doses of steroids >15mg/day for the last 3 months or with IV corticosteroids in the last 3 months
  * Patients under immunosuppressants for the last 3 months prior to recruitment with:

    * Methotrexate ≥25mg/week
    * Azathioprine ≥2.5mg/kg/day
    * Cyclosporine A > 3mg/kg/day
    * Mycophenolate Mofetil > 2gr/day
  * Treatment with cyclophosphamide (any dose or route of administration) or Belimumab in the past 6 months
  * Patients with combined therapy of two or more immunosuppressants
  * Patients on depletive therapy such as Rituximab in the last year
  * Patients receiving experimental therapy.
  * Chronic HBV or HCV infection
  * Overlap syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with systemic autoimmune diseases
Sampling Method: Probability Sample
Enrollment: 2006 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Gene expression in total blood | 2 years
  Gene expression will be done using commercial gene expression microarrays in total blood from all samples using the RNA Paxgene tube.
Flow cytometry analysis to determine cell proportions in the total blood mixture in all individuals. | 24 hours
  9 optimized panels of antibodies will be used to determine cell subpopulations in peripheral blood (including very minor cell populations).
Genotyping | 2 years
  Genotyping will be done using a whole genome array
Metabolite determination | 2 years
  Metabolite determination in plasma and urine using Nuclear Magnetic Resonance
Exosome isolation from plasma and urine | 2 years
  set up of the methodology for isolating exosomes in these bodily fluids for gene expression analysis
Cytokine profile determination | 2 years
  88 different cytokines will be assessed with Luminex
routine autoantibodies in serum | 2 years
  set of serum autoantibodies will be determined in a European validated laboratory. Also, they will perform detection of antibodies against small lipid moieties i.e.antiphosphorylcholine), lupus anticoagulant and complement proteins in plasma.
Gene methylation in total blood | 2 years
  Methylation analysis will be done using the methylome 450k array using the DNA obtained from total blood. MicroRNA gene expression arrays using total blood.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Alarcon, Study Director — Fundación Pública Andaluza Progreso y Salud (PHFSpain)
Locations (18):
- Medical University of Vienna, Vienna, Austria
- Belgium (2):
  - Université catholique de Louvain - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven - KU Leuven, Department of Rheumatology (KU LEUVEN), Leuven
- CHRU de Brest, Brest, France
- Germany (3):
  - Deutsches Rheuma-Forschungszentrum Berlin (DRFZ), Berlin
  - University of Cologne, Cologne
  - Medizinische Hochschule Hannover, Hanover
- University of Szeged, Szeged, Hungary
- Italy (2):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico (IRCCS), Milan
  - UNIMI, Istituto Ortopedico Getano Pini, Milan
- Centro Hospitalar do Porto, Porto, Portugal
- Spain (6):
  - Hospital Clinic I Provicia- Institut d'Investigacions Biomèdiques August Pi i Sunyer (IDIBAPS), Barcelona
  - Hospital Universitario Reina Sofía Andaluz de Salud, Córdoba
  - Hospital Universitario San Cecilio Servicio Andaluz de Salud, Granada
  - Hospital Virgen de las Nieves Granada, Granada
  - Hospital Regional de Málaga Servicio Andaluz de Salud, Málaga
  - Hospital Universitario Marqués de Valdecilla, Servicio Cántabro de Salud, Santander
- Hospitaux Universitaires de Géneve, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided